CLINICAL TRIAL: NCT06231446
Title: A Multicenter Prospective Cohort Study of the Clinical Characteristics and Prognosis of Respiratory Failure Patients With ECMO Therapy
Brief Title: Extracorporeal Membrane Oxygenation for Respiratory Failure Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Qingyuan Zhan, prof., China-Japan Friendship Hospital
Other Study IDs: 2022-KY-113-1
Record Dates: First submitted 2024-01-18; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Respiratory Failure Patients Treated With ECMO

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — This was an observational cohort study with no intervention for all enrolled patients.

SUMMARY:
The present study is a multicentre cohort study. Respiratory failure patients treated with extracorporeal membrane oxygenation (ECMO) were enrolled. Clinical data before and during ECMO treatment were collected. Clinical data before and during ECMO treatment were collected. By this retrospective clinical data and prospective study, to observe the current status of respiratory failure patients treated with ECMO in China, analyze the clinical characteristics and prognosis of patients, and explore the clinical prevention and treatment strategies of major complications of ECMO.

DETAILED DESCRIPTION:
Extracorporeal membrane oxygenation (ECMO) is the ultimate life support for critically ill patients. However, ECMO was developed relatively late in China, and the large number of applications in the field of respiratory failure originated from the 2009 H1N1 influenza epidemic in China. Since then, the number of respiratory failure patients with ECMO has increased year by year. Nevertheless, there are still many problems about ECMO therapy for respiratory failure in China, mainly as follows:(1) Lack of real-world clinical data on ECMO. Most centers do not have their own databases, lack long-term follow-up, and are unable to establish a mature ECMO quality management system. (2) Lack of ECMO-related biological sample libraries. (3) Risk factors for major complications such as thrombosis and hemorrhage, ventilator-associated pneumonia, and bloodstream infections are still unclear. At present, most of the experience in the prevention and treatment of major complications of ECMO comes from foreign studies, and clinical studies have confirmed that the sensitivity and specificity of the currently commonly used biological indicators in the prediction and early warning of complications are not ideal. Therefore, there is an urgent need to carry out research on new biomarkers based on the establishment of clinical databases and biospecimen libraries. We retrospectively collected clinical data on respiratory failure patients treated with ECMO from June 2019 from five hospitals, and prospectively enrolled respiratory failure patients treated with ECMO from October 2022 from five hospitals. By this cohort study, to establish clinical databases and biospecimen libraries, and analyze the clinical characteristics and prognosis of patients, and explore the clinical prevention and treatment strategies of major complications of ECMO.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 80 years.
2. The patient or guardian voluntarily signs an informed consent form.
3. If one of the following conditions is met.

   * ARDS patients: lung-protective ventilation (Vt 6ml/kg, PEEP ≥ 10cm H2O) combined with recruitment maneuver, prone position ventilation, or high frequency oscillation ventilation with PaO2/FiO2<100 mmHg or P(A-a)O2>600 mmHg under pure oxygen inhalation; or respiratory rate>35 breaths/min, pH<7.2 and plateau pressure>30 cmH2O, with VV-ECMO adjuvant therapy.
   * Lung transplantation patients with ECMO support during perioperative period.
   * Asthma patients: under invasive mechanical ventilation support, platform pressure >35cmH2O concomitant with severe respiratory acidosis (pH<7.1), or unstable hemodynamics, perform VV-ECMO or ECCO2R adjuvant therapy if there is no contraindication to ECMO,
   * Chronic Obstructive Pulmonary Disease (COPD): to enable patients with severe COPD requiring invasive ventilation to avoid intubation, or to assist in evacuation of tracheal intubation, perform ECMO adjuvant therapy;.
   * Perioperative ECMO support for elective surgeries such as high-risk or complex tracheobronchial surgeries and high-risk or complex pneumonectomies; 6). Patients judged by the investigator to be eligible for this study, such as thoracic surgery patients with high perioperative risk and prophylactic use of ECMO for perioperative safety.

Exclusion Criteria:

1. Age < 18 years or > 80 years.
2. Duration of positive pressure ventilation with tracheal intubation for more than 7 days prior to admission.
3. Combination of severe irreversible end-stage disease, such as cancer, end-stage of the hepatocirrhosis, etc.
4. Irreversible multiorgan failure.
5. Combined cerebrovascular events such as severe cognitive impairment, cerebral haemorrhage or stroke occurring within 3 months.
6. Severe coagulopathies or bleeding disorders, or the presence of contraindications to anticoagulation, or inability to administer systemic anticoagulation.
7. Patients who are pregnant or breastfeeding.
8. Severe peripheral vascular disease or difficulty with ECMO placement.
9. With other untreatable end-stage disease.
10. Other inappropriate conditions for this study in the opinion of investigators

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Respiratory failure patients with ECMO in China-Japan Friendship Hospital, The First Affiliated Hospital of Anhui Medical University, The Second Affiliated Hospital, Zhejiang University School of Medicine and Jiangxi Provincial People's Hospital.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | 30 days

SECONDARY OUTCOMES:
Duration of mechanical ventilation | From the onset of endotracheal intubation to the withdrawal of endotracheal intubation or death，an average of 5 weeks.
ECMO duration | From the onset of ECMO to the withdrawal of ECMO or death, an average of 4 weeks.
Length of stay in ICU | From ICU admission to ICU discharge or death, an average of 8 weeks.
Systemic and localized bleeding | From ICU admission to discharge or death, , an average of 8 weeks.
Ventilator-associated pneumonia | From ECMO run to 48 hours after ECMO withdrawal, an average of 6 weeks.
Catheter-related bloodstream infection | From ECMO run to 48 hours after ECMO withdrawal, an average of 4 weeks.
ECMO-related thrombosis | From the onset of ECMO to one week after the withdrawal of ECMO or death, an average of 4 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No